CLINICAL TRIAL: NCT05287438
Title: Next Generation Sequencing Versus Traditional Cultures for Clinically Infected Penile Implants: Impact of Culture Identification on Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MicroGenDX (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MDX-002
Record Dates: First submitted 2022-03-02; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Penile Implantation; Infections
Keywords: next generation sequencing; penile prosthesis; infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Group A will receive results based on standard culture and Group B will receive results based on NGS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Culture (Active Comparator): Following local standard of care, treatment will be based on standard culture
  Interventions: Diagnostic Test: Standard Culture
- Group B - NGS (Experimental): Treatment will be based on NGS results reviewed by an infectious disease doctor
  Interventions: Diagnostic Test: Next-Generation DNA Sequencing

INTERVENTIONS:
Diagnostic Test: Next-Generation DNA Sequencing — NGS is a technique of microbiological sequencing, using 16s ribosomal RNA molecular identification has been implemented to detect bacteria and fungi present in the sample
  Other Names: NGS
  Arms: Group B - NGS
Diagnostic Test: Standard Culture — Standard of care culture and sensitivity
  Arms: Group A - Culture

SUMMARY:
Randomized prospective study to evaluate next generation sequencing (NGS) and standard-of-care culture for clinically infected penile implants and to compare outcomes with identification of microbes.

DETAILED DESCRIPTION:
Randomized prospective study to evaluate next generation sequencing (NGS) and standard-of-care culture for clinically infected penile implants and to compare outcomes with identification of microbes. Eligible subjects will undergo a baseline/screening visit at which time the following will be collected: demographics/history/known allergies to antibiotics, symptom scoring questionnaire. Drainage swabs OR needle aspiration will be collected for standard culture and PCR/NGS and empiric antibiotics will start.

Subjects will be randomized into the culture arm or the NGS arm. If randomized to NGS: central ID reviews result according to arm and offers recommendations. Physician will treat based on antibiotic recommendations (based on positive PCR/NGS or positive culture, if negative then empiric treatment will be continued) adjusted for patients contraindications and co-morbidities If randomized to the traditional culture arm: Physician will follow routine local standard of care.

A follow-up visit will occur within 10 days of starting empiric antibiotic therapy to collect symptoms scoring questionnaire. A 2nd and final visit will occur 6 months after baseline to collect similar data to the 1st follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male penile prosthesis patients
* Age range: 18-80
* Within 6 months of penile prosthesis surgery
* At least 1 of the following: Device part stuck to thinning skin, any drainage from the wound site, massive red and swollen genitalia parts, exposed penile prosthesis parts, draining open tract, draining hematoma

Exclusion Criteria:

* Transgender / neophallus
* Not able to communicate or follow up well, or non-compliant
* Less than 18 or more than 80 years old
* Active addiction
* Main issue is implant pain

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Device survival rates by calculating by incidence of implant freely mobile and working without tenderness | 2 years
  To determine if device survival rates outcomes are improved using NGS versus traditional culture
Patient satisfaction of penile prosthesis | 2 years
  Satisfaction is a 5-point descriptive scale in which subjects self-report that degree of satisfaction: high, mostly, fair, minimum, and none

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - WK Advanced Urology, Bossier City, Louisiana
  - Duke University, Raleigh, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with other researchers

REFERENCES:
- [Background] Carrasquillo RJ, Munarriz RM, Gross MS. Infection Prevention Considerations for Complex Penile Prosthesis Recipients. Curr Urol Rep. 2019 Feb 1;20(3):12. doi: 10.1007/s11934-019-0875-7. PMID 30707308
- [Background] Krzastek SC, Smith R. An update on the best approaches to prevent complications in penile prosthesis recipients. Ther Adv Urol. 2019 Jan 8;11:1756287218818076. doi: 10.1177/1756287218818076. eCollection 2019 Jan-Dec. PMID 30671142
- [Background] Carvajal A, Benavides J, Garcia-Perdomo HA, Henry GD. Risk factors associated with penile prosthesis infection: systematic review and meta-analysis. Int J Impot Res. 2020 Nov;32(6):587-597. doi: 10.1038/s41443-020-0232-x. Epub 2020 Feb 3. PMID 32015525
- [Background] Mahon J, Dornbier R, Wegrzyn G, Faraday MM, Sadeghi-Nejad H, Hakim L, McVary KT. Infectious Adverse Events Following the Placement of a Penile Prosthesis: A Systematic Review. Sex Med Rev. 2020 Apr;8(2):348-354. doi: 10.1016/j.sxmr.2019.07.005. Epub 2019 Sep 10. PMID 31519461
- [Background] Carrasquillo RJ, Gross MS. Infection Prevention Strategies Prior to Penile Implant Surgery. Eur Urol Focus. 2018 Apr;4(3):317-320. doi: 10.1016/j.euf.2018.07.002. Epub 2018 Jul 13. PMID 30017899
- [Background] Levy PY, Fenollar F. The role of molecular diagnostics in implant-associated bone and joint infection. Clin Microbiol Infect. 2012 Dec;18(12):1168-75. doi: 10.1111/1469-0691.12020. PMID 23148447
- [Background] Salimnia H, Fairfax MR, Lephart PR, Schreckenberger P, DesJarlais SM, Johnson JK, Robinson G, Carroll KC, Greer A, Morgan M, Chan R, Loeffelholz M, Valencia-Shelton F, Jenkins S, Schuetz AN, Daly JA, Barney T, Hemmert A, Kanack KJ. Evaluation of the FilmArray Blood Culture Identification Panel: Results of a Multicenter Controlled Trial. J Clin Microbiol. 2016 Mar;54(3):687-98. doi: 10.1128/JCM.01679-15. Epub 2016 Jan 6. PMID 26739158
- [Background] Tzeng A, Tzeng TH, Vasdev S, Korth K, Healey T, Parvizi J, Saleh KJ. Treating periprosthetic joint infections as biofilms: key diagnosis and management strategies. Diagn Microbiol Infect Dis. 2015 Mar;81(3):192-200. doi: 10.1016/j.diagmicrobio.2014.08.018. Epub 2014 Nov 5. PMID 25586931